CLINICAL TRIAL: NCT00747981
Title: Management and Assessment of Thoracic CT Scan for Diagnosis of Aspirated Foreign Bodies in Children
Brief Title: Thoracic Computed Tomography Scan for Diagnosis of Aspirated Foreign Bodies.
Acronym: SICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: K 070601
Record Dates: First submitted 2008-09-05; First posted 2008-09-08 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Aspirated Foreign Body of Lower Respiratory Tract
Keywords: CT Scan; Endoscopy; Aspiration; Foreign Bodies
MeSH Terms: conditions — Foreign Bodies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Thoracic CT Scan
  Interventions: Procedure: Thoracic CT Scan

INTERVENTIONS:
Procedure: Thoracic CT Scan — Perform a CT Scan and an endoscopy

SUMMARY:
To access CT Scan as a diagnostic tool for foreign bodies aspiration.

DETAILED DESCRIPTION:
Comparison with gold standard diagnostic tool, the endoscopy

ELIGIBILITY:
Inclusion Criteria:

* age between 6 months and 16 years
* suspicion of a foreign body aspiration
* health care assurance
* information of parents

Exclusion Criteria:

* emergency situation
* certainly of foreign body presence
* delay for CT Scan realization longer than 24 hours
* no speaking French parents
* parents refusal.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 311 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Comparison between CT Scan and endoscopy results | 12 HOURS

SECONDARY OUTCOMES:
X Ray radiation induced by CT Scan | TWO YEARS

CONTACTS AND LOCATIONS:
Overall Officials: Yves MANACH, MD, HDR, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Paris V University & Assistance Publique Hôpitaux de Paris, Paris, France

REFERENCES:
- [Result] Manach Y, Pierrot S, Couloigner V, Ayari-Khalfallah S, Nicollas R, Venail F, Pondaven S, Baculard F, Tantcheu V. Diagnostic performance of multidetector computed tomography for foreign body aspiration in children. Int J Pediatr Otorhinolaryngol. 2013 May;77(5):808-12. doi: 10.1016/j.ijporl.2013.02.016. Epub 2013 Mar 13. PMID 23489882